CLINICAL TRIAL: NCT02091323
Title: Effect of Modified Laparoscopic Roux-en-Y Gastric Bypass Surgery on Type 2 Diabetics With Lower Body Mass Index in China
Brief Title: Effect of Laparoscopic Roux-en-Y Gastric Bypass Surgery on Non-severe Obesity With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Wu Liangping, chief, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Lrygb2014
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: T2DM, gastric bypass surgery, BMI<35, obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMI<28kg/m2 (Experimental): Indicators monitored preoperatively and at 1,3,6,12 months after surgery in BMI<28kg/m2 group.
  Interventions: Procedure: gastric bypass surgery
- control (Other): Indicators monitored preoperatively and at 1,3,6,12 months after surgery in BMI>28kg/m2 group as well.
  Interventions: Procedure: gastric bypass surgery

INTERVENTIONS:
Procedure: gastric bypass surgery — With the patient under intubation and general anesthesia, a pneumoperitoneum was created and the pressure was set to 15 mmHg. All LRYGB operations were performed using four trocars. Separate cardiac angle and hepatogastric ligament from the left gastric artery between 2 and 3 branch by hanging liver on the abdominal wall so as to enter into the lesser sac. Reveal the ligament of Treitz, lift the jejunum from the Treitz ligament 75 ~ 150 cm, connect the distal jejunum to the posterior wall of the stomach with a linear cutting staple by an end-to-side anastomosis and suture the common opening at last.
  Other Names: Roux-en-Y Gastric Bypass Surgery

SUMMARY:
The effect of roux-en-Y gastric bypass(RYGB) on patients with type 2 diabetes mellitus(T2DM) and a body mass index(BMI)>35kg/m2 is clear. There are large-scale patients with T2DM in Chinese population and currently about two-thirds of them are lack of adequate blood glucose control. Asian Chinese have different type of obesity, different style of diet, and a relatively low BMI levels as well. We assess the feasibility and efficacy of laparoscopic roux-en-Y gastric bypass surgery (LRYGB) in patients with non-severely obese T2DM.Taking into account the differences of body size and diet between the United States & Europe and Asian countries, diabetic situation has its special features in different regions, especially in Asia China. Asian Chinese have a high incidence of T2DM and a relatively low BMI levels. Evaluating the benefits from LRYGB for T2DM in Asian Chinese diabetes subjects with a body mass index of less than 35kg/m2 and looking for sufficient evidence to this operation become necessary.The patients will be followed up for one year after surgery and a comparison would be made between the two groups. Clinical indicators that reflect the effect of LRYGB are monitored before surgery and 1, 3,6,12 months after surgery. Complete remission of diabetes was defined by hemoglobin A1c (HbA1c)<6.0% and Fasting plasma glucose (FPG)<5.6mmol/L.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is well known as a chronic metabolic disease. As the main manifestation of T2DM , the disorder of glucose metabolism which is due to the gradual dysfunction of pancreatic islet and significant insulin resistance results in many problems and complications associated with T2DM such as hypertension, cardiovascular diseases(CVD), lipid disorders and other complications. Currently, there are more than 346 million people suffered from T2DM worldwide, among which T2DM accounts for about 90%. A report published by Chinese diabetes and metabolic syndrome research group in 2010 showed that overall prevalence of diabetes is 9.7% over the age of 20 and the total number of diabetes mellitus has reached 92.4 million in Chinese population and what's worse, more than 15.5 percent of adults are in the pre-diabetic state. Through traditional diet therapy, exercise, changing lifestyle, and standardized medical treatment have a certain effect on diabetes and its complications, T2DM can't be cured so far. How to cure diabetes mellitus and improve the quality of life of diabetic patients is a common problem faced by doctors in all countries. In 1984, Pories et al have found that glucose metabolism indicators significantly improved when he analyzed a report of three-year progress results of obesity patients with T2DM after laparoscopic Roux-en-Y gastric bypass surgery(LRYGB) , thus opening a door to the surgical treatment for diabetes. Now LRYGB is often performed in Europe and United State, and has been written into the diabetes treatment guidelines by American Diabetes Association in 2009. The surgical treatment for diabetes is an extension from the surgical treatment for morbid obesity. So diabetes treatment guidelines in 2014 show that bariatric surgery may be considered for T2DM with a body mass index （BMI） >35 kg/m2, especially if diabetes or associated comorbidities are difficult to control with lifestyle and pharmacological therapy. However, it also mentioned that small trials have shown benefit in patients with type 2 diabetes mellitus and BMI 30-35 kg/m2 after bariatric surgery. But it still lacks sufficient evidence for patients with BMI below 30kg/m2. A survey conducted in Shanghai, China, showed that the prevalence of type 2 diabetes was 9.8%, while the prevalence of obesity was 4.3%.But in the United States, the incidence of type 2 diabetes was 10.9% and the obesity population defined by a BMI ≥30 kg/m2 may account for one third of the total population in 2009-2010. In addition, patients in Asian countries are mostly abdominal obesity compared with that of patients in the United States and Europe where have different type of obesity. Taking into account the differences of body size and diet between the United States & Europe and Asian countries, diabetic situation has its special features in different regions, especially in Asia China. Asian Chinese have a high incidence of T2DM and a relatively low BMI levels. Evaluating the benefits from LRYGB for T2DM in Asian Chinese diabetes subjects with a body mass index of less than 35kg/m2 and looking for sufficient evidence to this operation become necessary.

ELIGIBILITY:
Inclusion Criteria: In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose(PG) ≥200 mg/dL(11.1 mmol/L) or fasting plasma glucose (FPG) ≥ 7 .0 mmol / L or Two-hour PG ≥200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test(OGTT) or HbA1c > 6.5% .The study candidates were included if they had any of the following features:

* exclusion of type 1 diabetes mellitus(T1DM) ;
* BMI ≤ 35 kg/㎡ or waist circumference >90cm;
* duration of T2DM less than 15 years ;
* age ≤ 65 years ;
* islet functional reserve :fasting C-peptide (FC-P) normal or more , postprandial two-hour C-peptide response more than 2 times compared with a pre-dinner ;
* poor control of medical treatment ,glycated hemoglobin (HbA1c) ≥ 7 .0%;
* volunteer to accept LRYGB surgery and sign the consent

Exclusion Criteria:

* type 1 diabetes mellitus
* age >65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
fasting plasma glucose(FPG) | up to 36 months after surgery

SECONDARY OUTCOMES:
hemoglobin A1c (HbA1c) | HbA1c will be monitored preoperatively and at 1,3,6,12 ,24,36months after surgery

OTHER OUTCOMES:
weight loss | weight loss will be monitored preoperatively and at 1,3,6,12,24,36 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Wu, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Cotillard A, Poitou C, Duchateau-Nguyen G, Aron-Wisnewsky J, Bouillot JL, Schindler T, Clement K. Type 2 Diabetes Remission After Gastric Bypass: What Is the Best Prediction Tool for Clinicians? Obes Surg. 2015 Jul;25(7):1128-32. doi: 10.1007/s11695-014-1511-8. PMID 25387683
- [Background] Luger M, Kruschitz R, Langer F, Prager G, Walker M, Marculescu R, Hoppichler F, Schindler K, Ludvik B. Effects of omega-loop gastric bypass on vitamin D and bone metabolism in morbidly obese bariatric patients. Obes Surg. 2015 Jun;25(6):1056-62. doi: 10.1007/s11695-014-1492-7. PMID 25381120
- [Background] Torriani M, Oliveira AL, Azevedo DC, Bredella MA, Yu EW. Effects of Roux-en-Y gastric bypass surgery on visceral and subcutaneous fat density by computed tomography. Obes Surg. 2015 Feb;25(2):381-5. doi: 10.1007/s11695-014-1485-6. PMID 25381117
- [Result] Chen Y, Zeng G, Tan J, Tang J, Ma J, Rao B. Impact of roux-en Y gastric bypass surgery on prognostic factors of type 2 diabetes mellitus: meta-analysis and systematic review. Diabetes Metab Res Rev. 2015 Oct;31(7):653-62. doi: 10.1002/dmrr.2622. Epub 2014 Dec 17. PMID 25387821